CLINICAL TRIAL: NCT03267485
Title: Expression of TET1 Gene in Acute Leukaemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Monica Botros Mosaad, Resident doctor of clinical pathology department South Egypt Cancer Institute, Assiut University
Other Study IDs: TET1 gene in acute leukemia
Record Dates: First submitted 2017-08-29; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Acute Leukemia
MeSH Terms: interventions — Real-Time Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: real time PCR — Real Time PCR is based on the detection of the fluorescence produced by a reporter molecule which increases, as the reaction proceeds. These fluorescent reporter molecules include dyes that bind to the double-stranded DNA or sequence specific probes . Moreover, there is no need for the post PCR processing which saves the resources and the time. .

SUMMARY:
The aim of the present study is to detect the expression of TET 1 gene in patients with acute leukemia and its correlation with clinical and pathological criteria of the patients.

DETAILED DESCRIPTION:
"Acute leukemia" is defined by the World Health organization standards, in which greater than 20% of the cells in the bone marrow are blasts (Kabuto et al., 2006). Cure is a realistic goal and is achieved in more than 80% of affected children, although only 20-40% of adults are cured(Rose-Inman and Kuehl, 2014).

There are two major forms of acute leukaemias-acute lymphoblastic leukaemia (ALL) and acute myeloid leukaemia (AML) Acute lymphoblastic leukemia (ALL) is an acute form of leukemiacharacterized by the overproduction and accumulation of cancerous, immature white blood cells, known as lymphoblasts(Rose-Inman and Kuehl, 2014).

Internationally, ALL is more common in Caucasians than in Africans; it is more common in Hispanics and in Latin America(Greer, 2014; Urayama and Manabe, 2014).About 6,000 cases are reported in the United States every year(Inaba et al., 2013).

Acute Myeloid leukemia (AML)Acute Myeloid Leukemia is a cancer of leukemic stem cells (LSCs) with a rapid progression. It is characterized by overproduction of immature myeloid cells in bone marrow which crowds out normal hematopoietic stem cells (HSC) (Indian J Hematol Blood Transfus. 2017).

DNA methylation is a covalent modification that is critical for the regulation of gene expression in a wide variety of biological contexts (Jaenisch and Bird, 2003; Bergman and Cedar, 2013). Methylation of DNA on cytosines is an important mechanism for silencing gene expression, and cytosine demethylation is required for gene activation (Ito et al., 2011; He et al., 2011). DNA methylation plays important roles in a variety of cellular processes, including genomic imprinting , X-chromosome inactivation and regulation of gene expression (Bird 2002).

The ten-eleven translocation (Tet) family of methylcytosine dioxygenases, which includes Tet1, Tet2, and Tet3 enzymes, has been recently implicated in DNA demethylation it converts 5-methylcytosine (5mC) to 5-hydroxymethylcytosine (5hmC) as well as to 5-formylcytosine and 5-carboxylcytosine (Tahiliani et al., 2009; Ito et al., 2010; Guo et al., 2011a). 5hmC has been proposed to act as an intermediate in demethylation and the base-excision repair machinery (Guo et al., 2011a).

Tet proteins contain several conserved domains (Tahiliani et al. 2009), including a CXXC domain that has high affinity for clustered unmethylated CpG dinucleotides and a catalytic domain that is typical of Fe(II)- and 2-oxoglutarate (2OG)-dependent dioxygenases (Loenarz and Schofield 2011) ), mutation of iron-binding sites of Tet proteins abolishes their enzymatic activities (Tahiliani et al. 2009; Ito et al. 2010). In addition, 2-hydroxyglutarate (2-HG), a competitive inhibitor of 2OG-dependent dioxygenases, suppresses the catalytic activity of Tet proteins (W Xu et al. 2011).Both fully methylated and hemimethylated DNA in a CG or non-CG context can serve as substrates for TET1 (Tahiliani et al. 2009; Ficz et al. 2011; Pastor et al. 2011). In tumor cells, the normal pattern of DNA methylation is often altered, resulting in global hypomethylation of the genome in conjunction with hypermethylation at CpG islands within the promoters of critical genes such as tumor suppressors (Esteller, 2008).

The TET1 gene, was initially identified in acute myeloid leukemia (AML) as a fusion partner of the histone H3 Lys 4 (H3K4) methyltransferase MLL (mixed-lineage leukemia) (Ono et al. 2002; Lorsbach et al. 2003). TET1 is significantly upregulated and plays an oncogenic role in MLL-rearranged leukemia, rendering TET1 as a potential target for treating this form of hematopoietic malignancy ( Huang et al., 2013). Tet1 is abundantly expressed in hematopoietic stem/progenitor cells (HSC/HPCs) and differentiated lineages such as B cells and myeloid cells (Huang et al., 2013; Li et al., 2011 ; Moran-Crusio et al., 2011)

ELIGIBILITY:
Inclusion Criteria:

- sample from acute leukemia patients at diagnosis or relapse . healthy subjects as control .

Exclusion Criteria:

* Patients having any other haematological malignancies.
* Patient with acute leukemia in remission

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: acute leukemia patients at diagnosis or relapse .
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
expression of TET1 gene in acute leukemia | baseline
  role of TET1 gene expression in leukemogenesis

REFERENCES:
- [Background] Jain A, Varma S, Garg R, Malhotra P. Unilateral Gynaecomastia in a Young Man with Chronic Myeloid Leukemia. Indian J Hematol Blood Transfus. 2017 Sep;33(3):448-450. doi: 10.1007/s12288-016-0762-z. Epub 2016 Dec 19. PMID 28824259
- [Background] Lee BS, Jan YD, Huang GS, Huang CH, Chou HY, Wang JS, Tseng WY. Effect of dentin bonding agent diffusing through dentin slices on the reactive oxygen species production and apoptosis of pulpal cells. J Formos Med Assoc. 2015 Apr;114(4):339-46. doi: 10.1016/j.jfma.2012.12.009. Epub 2013 Feb 13. PMID 25839767